CLINICAL TRIAL: NCT05708378
Title: Comparison of Rocker Board and Stable Surface Training on Postural Stability, Balance and Gait in Stroke
Brief Title: Comparison of Rocker Board and Stable Surface Training on Postural Stability, Balance and Gait
Acronym: ACAMCAOAMMSE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/01489 Zarafshann
Record Dates: First submitted 2023-01-22; First posted 2023-02-01 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Stroke
Keywords: Rocker board training, postural stability, balance, gait
MeSH Terms: conditions — Stroke | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: participants and outcome assessors will be kept blinded about the intervention which the patients will be going to receive
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rocker board training (Experimental): Stretching Exercises (Heel drop, heel raises, Hamstring stretch, quad stretch, half kneel, IT band stretch, half squats). Hold the stretch for 20 seconds and repeat 10 times.
  Isometric Strengthening Exercises of calves, hamstrings, quads, hip flexors, gluteus, dorsiflexors and plantarflexors. Hold for 20 seconds and repeat 10 times.
  Pelvic Bridging Exercises. Trunk control exercises on Rocker Board in standing position first in medio-lateral direction for 10 min and then in anterio-posterior direction for 10 min with breaks in between.
  Interventions: Other: Rocker board training
- Stable surface training (Other): Stretching Exercises (Heel drop, heel raises, Hamstring stretch, quad stretch, half kneel, IT band stretch, half squats). Hold the stretch for 20 seconds and repeat 10 times.
  Strengthening Exercises calves, hamstrings, quads, hip flexors, gluteus, dorsiflexors and plantarflexors. Hold for 20 seconds and repeat 10 times.
  Pelvic Bridging Exercises. Trunk balance exercise (flexion, extension of lower and upper trunk, rotation of lower and upper trunk, forward and lateral reach) on plain surface.
  Interventions: Other: Stable surface training

INTERVENTIONS:
Other: Rocker board training — Patients will perform 24 sessions (4 times per week over 6 weeks) and effects will be measured before treatment, at 3rd and after 6th week.
  Other Names: Experimental group
  Arms: Rocker board training
Other: Stable surface training — Patients will perform 24 sessions (4 times per week over 6 weeks) and effects will be measured before treatment, at 3rd and after 6th week.
  Other Names: Control group
  Arms: Stable surface training

SUMMARY:
There is limited literature for the evaluation of comparison between effectiveness of postural control and balance training program on stable surface and unstable surface. So this study will help to improve reactive postural control in stroke patients which ultimately improve their walking capability, mobility and level of independence. This study will also enable the individual to be more independent and minimize their falls.

DETAILED DESCRIPTION:
Stroke is the second cause of death and the third cause of disability worldwide. It leads towards severe disability having a great impact upon independent activities of daily living. Postural stability and balance is often affected by strokes. Balance is a complex function with dynamic and static components. It is a major determinant of community ambulation and gait performance following strokes. Falls in post-stroke patients commonly occur due to impairment of balance. Hence, one of the primary objectives in stroke rehabilitation is to restore postural stability and functional balance, which is a combination of dynamic, static and reactive balance. For improving postural stability and balance one such technique is the utilization of a rocker board, where a platform positioned on an unstable surface is used to challenge balance. Whilst rocker boards have been used effectively for, postural stability, injury prevention, rehabilitation and balance enhancement. Improvements in rocker board performance may be attributable to one or more of the following: muscle strengthening, enhanced intersegmental coordination, increase in brain activity in the supplementary motor area and/or enhanced feed-forward and feed-backward postural control mechanisms. Postural instability limits lower limb functional activities, hence; rapid and optimal improvement of postural control in stroke patients is essential for their independence, social participation and general health. Improvement in postural stability have a great impact upon balance and gait. Rocker board training is also effective for gait and trunk balance in stroke patients. Postural stability increases due to unstable surface because perturbations felt by patients and consequent trails to compensate while doing exercises on the tilted Rocker Board activate the motor system of the patients. Neural plasticity may be enhanced by regular and repeated administration of this training. The trunk exercises on an unstable surface sensitize the muscle spindle through gamma motor neurons, thereby improving motor output which influences the stability of joint. Exercises on an unstable surface increases the external swing which more effectively encourages postural orientation by forcing faster modifications of the sensory and motor systems and also assists in the postural strategy of self-postural control. The trunk stabilization in stroke patients in an important prognostic factor of the recovery of balance ability and functional ambulation. The gait and balance improvement is because the motor cortex precedes from proximal to distal, the improved level of proximal trunk control leads to improvement in distal lower limb control which helped in altering better balance and gait. The relationship between postural control and improved mobility is already established. Through this study we want to improve postural stability through rocker based training and ultimately patient's dynamic balance and gait so functional capability of stroke patients can be enhanced.

ELIGIBILITY:
Inclusion Criteria:

* Both genders
* Age: between 40-60 years.
* Unilateral hemiplegia.
* ACA and MCA lesions only.
* Subacute and chronic stroke patients.
* First time affected.
* No visual and sensory deficits.
* Ambulatory stroke patients scoring 21 to 40 on Berg Balance Scale.
* Scoring > 21 on MMSE.

Exclusion Criteria:

* ● Any other neurological deficits as multiple sclerosis, Parkinsons disease etc.

  * Any musculoskeletal disorders like OA, ligament injury etc.
  * Non-ambulatory patients

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2023-06-10 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Beg Balance Scale | 6 weeks
  It is used to assess balance. , "Change will be measured from Baseline to 6 weeks"
Trunk Impairment Scale | 6 weeks
  It is used to measure motor impairment of the trunk after stroke. "Change will be measured from Baseline to 6 weeks"
Postural Assessment Scale for Stroke Patients | 6 weeks
  It is used for the assessments of postural control in stroke patients. "Change will be measured from Baseline to 6 weeks"
Timed Up and Go Test | 6 weeks
  It is for the assessment of lower extremity function, mobility and fall risk. "Change will be measured from Baseline to 6 weeks"
Functional Gait Assessment | 6 weeks
  It is for assessment of postural stability during walk. "Change will be measured from Baseline to 6 weeks"
Timed Walking Test | 6 weeks
  It is used for assessing functional status or fitness. "Change will be measured from Baseline to 6 weeks"

SECONDARY OUTCOMES:
Stroke Self-Efficacy Questionnaire | 6 weeks
  It evaluate self-efficacy as a result of being able to successfully perform a specific action in stroke patients. "Change will be measured from Baseline to 6 weeks"

CONTACTS AND LOCATIONS:
Overall Officials: Aruba Saeed, PhD*, Principal Investigator — Riphah International University Pakistan
Locations (1):
- Chinnar Hospital, Abbottabad, Khyber Pakhtunkhwa, Pakistan

IPD SHARING:
Plan to Share IPD: No